CLINICAL TRIAL: NCT06999512
Title: Impact of Comprehensive Geriatric Management on Morbidity and Quality of Life in Elderly Patients Undergoing Major Hepatectomy and Pancreaticoduodenectomy for Cancer. A Randomized Controlled Trial.
Brief Title: Impact of Comprehensive Geriatric Management on Morbidity and Quality of Life in Elderly Patients Undergoing Major Hepatectomy and Pancreaticoduodenectomy for Cancer
Acronym: HPB70+
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP230898; ID RCB (Other: 2024-A00038-39)
Record Dates: First submitted 2025-04-25; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hepatobiliary Cancer; Pancreatic Cancer
Keywords: patient over 70 years; hepatocellular carcinoma; intra-hepatic and peri-hilar cholangiocarcinoma; gallbladder cancer; peri-ampullary malignant tumors; pancreatic adenocarcinoma; colorectal liver metastases; Major Hepatectomy; Pancreaticoduodenectomy
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Hepatocellular; Gallbladder Neoplasms | interventions — Geriatric Assessment

STUDY DESIGN:
Intervention Model Description: prospective comparative randomized controlled open label multicentric trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): standard care follow up for the patient: Routine preoperative workup, routine postoperative follow-up
- Interventional group (Experimental): standard care follow up for the patient: Routine preoperative workup, routine postoperative follow-up with Perioperative geriatric management: CGA, preoperative geriatric consultation, perioperative tailored intervention, postoperative geriatric follow-up
  Interventions: Procedure: Comprehensive Geriatric Assessment

INTERVENTIONS:
Procedure: Comprehensive Geriatric Assessment — CGA:
  * Preoperative geriatric consultation
  * Perioperative tailored intervention if needed
  * Postoperative geriatric follow-up
  * M3 geriatric consultation
  Arms: Interventional group

SUMMARY:
The worldwide incidence of hepatobiliary and pancreatic (HPB) cancers is dramatically increasing especially for pancreatic cancer. Increasing age is associated with increased cancer risk. In North America and Europe, most people who are diagnosed with cancer every year are aged 65 years or older. Hepatectomy for hepatocellular carcinoma, intra hepatic and hilar cholangiocarcinoma, gallbladder cancer and hepatic metastases from colorectal cancer allows better survival compared to other treatments. Similarly, pancreaticoduodenectomy (PD) is the standard of care in patients with distal cholangiocarcinoma and patients with resectable pancreatic adenocarcinoma located in the head of the pancreas. This results in an increasing number of elderly patients being evaluated for hepatic and pancreatic surgery. Major hepatectomy and PD are amongst the most invasive and complex procedures in general surgery with high rates of morbidity as well as negative impact on quality of life. Many studies have reported poor post-surgical outcomes in the elderly patients, especially related to co-morbidities that characterizes this population such as, polypharmacy, cognitive decline, depression and malnutrition. The age in elderly cancer patient is not just a number. The management of these patients should not be limited to oncological care, but it should be extended to different clinical domains including physical, cognitive, psychological, socioeconomic and environmental aspects. In this population, the risk of adverse postoperative outcomes is not adequately described by routine format of current preoperative evaluation, such as age, comorbidities and other traditional tests. Furthermore, the Comprehensive Geriatric Assessment (CGA) is scarcely considered. The aim of CGA is to identify current health problems and to guide interventions thus reducing adverse outcomes and optimizing the functional status of older adults. Several trials have indeed shown that CGA and perioperative tailored interventions reduce morbidity and improve patient survival in other surgical disciplines. Similar data is lacking in both hepatic and pancreatic surgery.

The hypothesis is that CGA with perioperative tailored interventions could reduce postoperative morbidity in elderly patients after major hepatectomy and pancreaticoduodenectomy for cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 70 years, with histologically proven or clinical diagnosis of HPB cancer among the following:
* hepatocellular carcinoma
* intra-hepatic and peri-hilar cholangiocarcinoma
* gallbladder cancer
* peri-ampullary malignant tumors
* pancreatic adenocarcinoma
* colorectal liver metastases
* Needing one of the following procedures:
* Pancreaticoduodenectomy
* Major Hepatectomy (≥ 3 hepatic segments)

Exclusion Criteria:

* Patients who have no access to the French health system.
* Patient unable to sign informed consent.
* Patients included in a double-blind randomized trial
* Patients legally protected

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 526 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complex Index (CCI) value | 90 days after surgery
  Comparison of the 90-day postoperative morbidity between patients in the interventional arm (receiving preoperative CGA and perioperative tailored geriatric interventions) and those in the control arm (receiving standard of care).
  CCI is based on the Clavien-Dindo classification, and takes into account all cumulative complications and receives values between 0 (no complication) and 100 (death).

SECONDARY OUTCOMES:
Quality of life scale: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | at 3, 6 and 12 months post surgery
  Quality of life will be measured at the enrolment visit (baseline) and at 3, 6 and 12 months after surgery (M3, M6 and M12), using the EORTC QLQ-C30
Quality of life scale EQ-5D-5L | at 3, 6 and 12 months post surgery
  Quality of life will be measured at the enrolment visit (baseline) and at 3, 6 and 12 months after surgery (M3, M6 and M12), using the EQ-5D-5L
Quality of life scale ELD14 | at 3, 6 and 12 months post surgery
  Quality of life will be measured at the enrolment visit (baseline) and at 3, 6 and 12 months after surgery (M3, M6 and M12), using the ELD14.
Discharge status | 90 days after surgery
  Discharge status at 3 months after surgery (M3): home, rehabilitation facility, and still hospitalized or deceased
All-cause mortality at 90 days after surgery | at 3 months post surgery
  90-day postoperative mortality
complication occurence and classification | at 3 months post surgery
  Occurrence of all complications classified as grade II, III, IV, according to Clavien-Dindo scale within 90 days after surgery
Post-operative hospital length of stay (in days) | through study completion (an average of 5.5 years)
  Post-operative hospital length of stay (in days) defined as the time from surgery to the post-operative discharge date, transfer to a subacute service or death whichever comes first.
Post-operative ICU length of stay (in days) | through study completion (an average of 5.5 years)
  Post-operative ICU length stay (in days) defined as the time from the postoperative ICU entry date to ICU discharge date or death whichever comes first.
Loss of independence at 3 months after surgery | 90 days after surgery
  Loss of independence at 3 months after surgery (M3) defined by a score lower than 6/6 in ADL
Time (in days) between the date of randomization and the date of surgery | from randomization to surgery, a maximum of 1 month
  To compare between arms (interventional vs control arms) the delay between randomization and surgery
Overall survival | at 12 months post surgery
  Overall survival defined as the time from surgery to death from any cause over 1 year follow-up
time from surgery to cancer recurrence or death from any cause | through study completion (an average of 5.5 years)
  Disease-free survival defined as the time from surgery to cancer recurrence or death from any cause over 1 year follow-up
Percentage of patients that completed the geriatric intervention | through study completion (an average of 5.5 years)
  To estimate, within the interventional arm the proportion of patients who underwent the complete geriatric intervention
Percentage of patients contraindicated to surgery after CGA | through study completion (an average of 5.5 years)
  To estimate, within the interventional arm the proportion of patients definitively contraindicated to surgery after CGA because too frail
Time (in days) between the dates of randomization and preoperative geriatric consultation | through study completion (an average of 5.5 years)
  To estimate, within the interventional arm the delay between randomization and preoperative geriatric consultation
Time (in days) between the dates of preoperative geriatric consultation and onset of tailored interventions | through study completion (an average of 5.5 years)
  To estimate, within the interventional arm the delay between preoperative geriatric consultation and tailored interventions
Time (in days) between the dates of preoperative geriatric consultation and surgery | through study completion (an average of 5.5 years)
  To estimate, within the interventional arm the delay between preoperative geriatric consultation and surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella PITTAU, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (12):
- France (12):
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Chru Lille - Hopital Huriez, Lille
  - Hôpital Croix Rousse, HCL, Lyon
  - Hôpital Edouard Herriot, HCL, Lyon
  - Hôpital La Timone, Marseille
  - Hôpital Cochin, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU ROUEN - Site Charles Nicolle, Rouen
  - Hôpital Rangueil, Toulouse
  - Hôpital Paul-Brousse, Villejuif
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) collected in this study available.